CLINICAL TRIAL: NCT03996122
Title: Research of Anatomo-functional Biomarkers in Schizophrenia
Acronym: CLOZAREST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-A03281-54
Record Dates: First submitted 2019-05-23; First posted 2019-06-24 (Actual); Last update posted 2019-06-24 (Actual); Status verified 2019-06

CONDITIONS: Schizophrenia
Keywords: schizo-affective disorder; utra-resistance; clozapine; biomarker; fMRI
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — BDNF samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- resistant patients with schizophrenia: Age 18 - 60 years No MRI contraindication
  Interventions: Other: fMRI

INTERVENTIONS:
Other: fMRI — 3 fMRI (TO, Month 2 and Month 6) 3 BDNF samples (TO, Month 2 and Month 6)
  Other Names: BDNF samples

SUMMARY:
To objectify UR biomarkers, we propose a longitudinal follow-up of resistant patients with schizophrenia, starting before the onset of clozapine and including a multimodal brain imaging assessment (T1 and T2 weighted sequences, DTI, ASL-Perfusion, fMRI- Rest) associated with clinical and biological monitoring. In order to correct the MRI signal of clozapine hemodynamic effects, we will develop a new MRI methodology based on the concomitant collection of physiological parameters (blood pressure, electrocardiogram and respiration).

DETAILED DESCRIPTION:
The identification of biomarkers of ultra-resistance (UR) to treatment in schizophrenia would allow earlier, better adapted and more effective personalized management of these patients, which would improve their functional prognosis.

An early decrease in functional connectivity (FC) between some rest networks has recently been proposed as an UR biomarker by McNabb et al. Nevertheless, clozapine has, among its side effects, a direct cardiac action that profoundly modifies patient's hemodynamics. However, functional brain imaging techniques are based on BOLD effect which is dependent on these hemodynamic parameters. It is therefore not possible to say whether these differences in FC are inherent to the pathology or whether they are related to clozapine instauration which causes hemodynamic changes that may disturb BOLD signal.

To objectify UR biomarkers, investigators propose a longitudinal follow-up of resistant patients, starting before clozapine instauration and including a multimodal brain imaging assessment (T1 and T2 weighted sequences, DTI, ASL-Perfusion, fMRI- Rest) associated with clinical and biological monitoring. In order to correct the MRI signal of clozapine hemodynamic effects, investigators will develop a new MRI methodology based on the concomitant collection of physiological parameters (blood pressure, electrocardiogram and respiration).

ELIGIBILITY:
Inclusion Criteria:

* schizophrenia or schizoaffective disorder (DSM 5)
* drug resistance
* written patient approval
* social security number in France
* curator or tutor approval if needed

Exclusion Criteria:

* pregnancy
* other research participation
* neurological evolution disorder
* no MRI contraindication

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: resistant schizophrenia or schizoaffective disorder patients
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2019-04-04 (Actual); Primary Completion 2021-04-04 (Estimated); Study Completion 2021-10-04 (Estimated)

PRIMARY OUTCOMES:
functional resonance imaging: resting-state | baseline, Month 2 and Month 6
  Functional connectivity comparison between baseline, month 2 and month 6

SECONDARY OUTCOMES:
BDNF samples | baseline, Month 2 and Month 6
  BDNF concentration comparison between baseline, month 2 and month 6
functional resonance imaging: ASL | baseline, Month 2 and Month 6
  Cerebral perfusion comparison between baseline, month 2 and month 6
anatomical resonance imaging: DTI | baseline, Month 2 and Month 6
  Anatomical connectivity comparison between baseline, month 2 and month 6
anatomical resonance imaging: T1 | baseline, Month 2 and Month 6
  White and gray matter volumetric comparison between baseline, month 2 and month 6

CONTACTS AND LOCATIONS:
Overall Officials: Anaïs Vandevelde, MD, Principal Investigator — CHU of Caen, Esquirol
Locations (1):
- CHU CAEN Normandie, Caen, Normandy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Abnormalities of fronto-subcortical pathways in schizophrenia and the differential impacts of antipsychotic treatment: a DTI-based tractography study — https://www.ncbi.nlm.nih.gov/pubmed/30145382
- See also: Functional network dysconnectivity as a biomarker of treatment resistance in schizophrenia — https://www.ncbi.nlm.nih.gov/pubmed/29042073